CLINICAL TRIAL: NCT01267409
Title: Mapping and Manipulating the Emotional Territories of the Subthalamic (STN) Area in Deep Brain Stimulation (DBS) Treated Parkinson Patients
Brief Title: Mapping and Manipulating the Emotional Territories of the Basal Ganglia in PD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Renana Eitan, Dr, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EmotionalPD-HMO-CTIL
Record Dates: First submitted 2010-12-21; First posted 2010-12-28 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease
Keywords: Mapping the emotional territories of the STN; Identifying the emotional spectral signature of the STN single unit activity; Manipulating emotional processing of PD patients by high and low frequency stimulation; Affecting long-term emotional states of the PD patients
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: STN stimulation — Manipulating emotional processing of PD patients by high and low frequency stimulation of their subthalamic area (through the 4 DBS contacts) after the surgery

SUMMARY:
Depressive symptoms of Parkinson's disease (PD) patients are major predictors of their prognosis and quality of life. Using subthalamic nucleus (STN) deep brain stimulation (DBS) as an antidepressant could be a promising new direction. Existing methods of adjustment of DBS parameters aim at amelioration of the motor signs and therefore with inactivation of the STN motor territory only. Although the DBS parameter setting is believed to influence the mental state, there is no data that correlates stimulation parameters with mental state. The investigators hypothesize that the emotional territories of the STN have distinct electrophysiological properties and that specific stimulation of these emotional territories can influence the mental state and thus treatment with emotionally-adjusted DBS can improve the psychiatric symptoms of PD. In this project, the investigators intend to map the emotional territories of the STN using neuronal (single units) responses to emotional voices and to identify the emotional spectral signature of the STN single unit activity using spectral analysis and neuronal responses to emotional voices. The investigators also intend to investigate the emotional processing of PD patients by manipulating the stimulation of the subthalamic area. The proposed study will combine neural recording, stimulation and psychological tests to shed new light on emotional processing in the basal ganglia, as well as to provide better treatment for PD emotional disorders,

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite PD treated / candidates for treatment with DBS (patients with advanced idiopathic PD who are deemed appropriate for DBS surgery).
2. Patients will be included in the study irrespective of whether a diagnosis of major depression (MDD) (mild to moderate but not severe MDD) is fulfilled at baseline. Patients without depression will be monitored in the study for evidence of treatment emergent depression. Patients with depression will be monitored for antidepressant effects of stimulation change.
3. Age 40-75 years
4. Male or female.
5. Competent and willing to give written informed consent

Exclusion Criteria:

1. Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2].
2. Comorbidity with any Psychotic Disorder, Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Eating Disorder.
3. Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months
4. Significant cognitive decline, as measured by Addenbrooke's Cognitive Examination (ACE) and the Frontal Assessment Battery (FAB).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological recording and STN mapping | 24 m
  Mapping the emotional territories of the STN using neuronal (single units) responses to emotional voices during surgery.
  Manipulating emotional processing of PD patients by high and low frequency stimulation of their subthalamic area during and after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Renana Eitan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel